CLINICAL TRIAL: NCT03327844
Title: Regenerative Endodontic Therapy (RET) Using Antibiotic Pastes or Calcium Hydroxide Disinfection for the Management of Immature Non-vital Permanent Teeth in Children: A Randomized Controlled Clinical Trial
Brief Title: Regenerative Endodontic Therapy (RET) for the Management of Immature Non-vital Permanent Teeth in Children
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National University Health System, Singapore (Other)
Collaborators: National University of Singapore (Other); Health Promotion Board, Singapore (Other Government)
Responsible Party: Principal Investigator, Tong Huei Jinn, Consultant, National University Health System, Singapore
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DSRB 2015/00612
Record Dates: First submitted 2017-10-05; First posted 2017-11-01 (Actual); Last update posted 2021-10-21 (Actual); Status verified 2021-10

CONDITIONS: Infected Immature Permanent Teeth
Keywords: Regenerative Endodontic Therapy; Infected immature permanent teeth
MeSH Terms: interventions — Ciprofloxacin; Metronidazole; Calcium Hydroxide

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RET using bi-Antibiotics (Active Comparator): Interventions: Bi-antibiotics (Ciprofloxacin and Metronidazole) placed into the root canal during first treatment stage (disinfection stage)
  Interventions: Drug: RET using antibiotics (Ciprofloxacin and Metronidazole)
- RET using non-setting Calcium Hydroxide (Active Comparator): Interventions: non-setting calcium hydroxide placed into the root canal during first treatment stage (disinfection stage)
  Interventions: Drug: RET using non-setting Calcium Hydroxide

INTERVENTIONS:
Drug: RET using antibiotics (Ciprofloxacin and Metronidazole) — RET using antibiotics Ciprofloxacin and Metronidazole. First Treatment Visit: Local analgesic, tooth isolation, access, pulp extirpation and root canal irrigation with 1.5% sodium hypochlorite. Canal drying using paper points. Delivery of mixture of Bi antibiotic paste (Ciprofloxacin and Metronidazole with sterile water). Tooth access sealed with temporary dressing. Second Treatment Visit: Tooth analgesia using plain local analgesics without vasoconstriction, isolation and re-access as described above. Irrigation of root canal system using sodium hypochlorite followed by paper point drying. Initiation of bleeding through insertion of a sterile k-file at a length of 2-3 mm beyond the working length into the periapical tissues. Access sealed using resorbable plug, Biodentine, followed by composite resin.
  Other Names: Bi-Antibiotics
  Arms: RET using bi-Antibiotics
Drug: RET using non-setting Calcium Hydroxide — First Treatment Visit: Local analgesic, Tooth isolation, access, pulp extirpation and root canal irrigation with 1.5% sodium hypochlorite. Canal negotiation, canal drying using paper points. Delivery of the non-setting Calcium Hydroxide. Tooth access sealed with temporary dressing. Second Treatment Visit: Tooth analgesia using plain local analgesics without vasoconstrictor, isolation and re-access as described above. Irrigation of root canal system using sodium hypochlorite followed by paper point drying. Initiation of bleeding through insertion of a sterile k-file at a length of 2-3 mm beyond the working length into the periapical tissues. Access sealed using resorbable plug, Biodentine, followed by composite resin.
  Other Names: Calcium hydroxide
  Arms: RET using non-setting Calcium Hydroxide

SUMMARY:
This study evaluates the efficacy of Antibiotic pastes or Calcium hydroxide disinfection on healing of periapical pathology and continued root development of infected non-vital immature permanent teeth in children.

In the test group regenerative endodontic therapy (RET) is performed with antibiotics as the disinfecting agent, in the control group RET is performed with Calcium Hydroxide as the disinfecting agent.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 6-16 years of age
2. Patients who are fit and healthy or with American Society of Anesthesiologists (ASA) 1 or ASA 2 medical conditions
3. Patients with cooperation level that would allow treatment under local analgesia, application of rubber dam isolation and taking of intraoral radiographs.
4. Patients with permanent premolars that have incomplete root formation with an open apex of greater than 1mm width as observed radiographically and of single root canal morphology (22)
5. Patients with single rooted immature permanent premolars having one of the following pulpal and periapical diagnosis:

   a. Pulpal i. Necrotic pulp ii. Symptomatic and inflamed pulp not expected to heal. During attempted Cvek or cervical pulpotomy procedures, if the pulpal bleeding does not stop with direct pressure within 5 minutes, pulpectomy will be carried out and the patient will be recruited for RET procedures.

   b. Periapical i. Symptomatic apical periodontitis (with or without a radiographic apical lesion) ii. Asymptomatic apical periodontitis (with a radiographic apical lesion) iii. Acute apical abscess iv. Chronic apical abscess Teeth will be deemed non-vital if either are non-responsive to sensibility tests (i.e. Electric Pulp test and cold tests), and/or present with signs and symptoms of non-vitality (e.g. swelling and abscess).

Exclusion Criteria:

1. Patients aged > 16 years of age.
2. Patient with known allergies to Ciprofloxacin (or any fluoroquinolones class of antibiotics) or metronidazole antibiotics.
3. Patients with medical conditions and/or receiving medications that would affect:

   1. Their body's ability to heal e.g. Diabetes; or
   2. Their ability to clot efficiently, e.g. Haemophilia
4. Patients with risk of developing infective endocarditis or immune compromised patients.
5. Patients with non-vital permanent premolars where root development is already deemed to be completed (i.e. foramen size of 0-1.0mm diameter as determined radiographically).
6. Impacted or horizontally tilted teeth.
7. Concurrent signs of irreversible pathological root resorption determined radiographically, e.g replacement or internal root resorption, which could otherwise affect the prognosis of the tooth.
8. Uncooperative patients, or those unable to cope with treatment under local anaesthesia, rubber dam isolation and taking of intraoral radiographs.

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2021-07-31 (Actual)

PRIMARY OUTCOMES:
Resolution periapical radiolucency (Clinical evaluation) | 18 months (reviews are at periodicity of 3 months)
  Clinical evaluation: Presence/Absence of clinical signs of pain and soft tissue pathology (e.g. abscess, sinus tract etc.)
Resolution periapical radiolucency (Radiographic evaluation) | 18 months (reviews are at periodicity of 3 months)
  Size of periapical lesion will be graded using Periapical Index (PAI)

SECONDARY OUTCOMES:
Continued root development (Radiographic evaluation) | 18 months (reviews are at periodicity of 3 months)
  Quantitative outcomes of lengths and thickness will be measured in millimeters (mm).
Discolouration of tooth | 18 months (reviews are at periodicity of 3 months)
  Changes in tooth colour will be measured through assessment of photographs
Patient reported outcomes (Perceived oral health-related quality of life (OHRQL)) | 18 months (reviews are at periodicity of 3 months)
  Oral health related quality of life will be evaluated using the validated questionnaire Child-Oral Impacts on daily performances (C-OIDP)
Patient reported outcomes (Quantitative pain rating) | 18 months (reviews are at periodicity of 3 months)
  Quantitative pain rating will be done using Faces Pain scale for children 12 years and below; and Numeric Rating scale (NRS) for children 13 years and above.
  Faces Pain Scale (range: 0-10); higher scores indicate worse pain
  Numeric Rating scale (range: 0-10; 0 - no pain, 1-3 - mild pain, 4-6 - moderate pain, 7-10 - severe pain); higher scores indicate worse pain

CONTACTS AND LOCATIONS:
Overall Officials: Huei Jinn Tong, Principal Investigator — National University Health System
Locations (2):
- Singapore (2):
  - School Dental Service, Health Promotion Board, Singapore
  - National University Hospital, Singapore

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol (2017-08-21): https://cdn.clinicaltrials.gov/large-docs/44/NCT03327844/Prot_000.pdf
  • Informed Consent Form (2017-02-17): https://cdn.clinicaltrials.gov/large-docs/44/NCT03327844/ICF_001.pdf